CLINICAL TRIAL: NCT02730611
Title: The Influence of Metabolic Syndrome and Circulating Bile Acid Levels on the Development of Hepatocellular Carcinoma and Biliary Tract Cancers
Brief Title: Metabolic Syndrome, Bile Acids, Hepatocellular Carcinoma and Cholangiocarcinoma
Acronym: METSLIVER
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Centre International de la Recherche sur le Cancer (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PRT-K14-038
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Morbid Obesity; Vertical Sleeve Gastrectomy; Metabolic Syndrome; Hepatocellular Carcinoma; Cholangiocarcinoma; Disorder of Bile Acid and Cholesterol Metabolism
Keywords: Vertical sleeve gastrectomy; Metabolic syndrome; Disorder of Bile Acid and Cholesterol Metabolism; Cholangiocarcinoma; Hepatocellular carcinoma
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces, blood, liver biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with morbid obesity and vertical sleeve gastrectomy

SUMMARY:
Increasing rates of highly malignant hepatocellular carcinoma (HCC) and biliary tract cancers (GBTC) observed in Western populations may be related to obesogenic lifestyle factors and their metabolic consequences, such as metabolic syndrome (MetS), inflammation and altered production of bile acids (BA). Such lifestyle behaviours may induce changes in the gut microflora which in turn affect BA profiles, increasing their carcinogenicity. Some elevated BA may be oncogenic in exposed liver, bile ducts and gall bladder. Vertical sleeve gastrectomy may change bile acid composition.

The aims of this study are:

1. whether specific presurgical bila acid profiles are predictive of efficacy of vertical sleeve gastrectomy, reflective of liver function and metabolic dysfunction;
2. whether specific presurgical bile acid profiles are predictive of the efficacy of sleeve gastrectomy

DETAILED DESCRIPTION:
"Increasing rates of highly malignant hepatocellular carcinoma (HCC) and biliary tract cancers (GBTC) observed in Western populations may be related to obesogenic lifestyle factors and their metabolic consequences, such as metabolic syndrome (MetS), inflammation and altered production of bile acids (BA). Such lifestyle behaviours may induce changes in the gut microflora which in turn affect BA profiles, increasing their carcinogenicity. Some elevated BA may be oncogenic in exposed liver, bile ducts and gall bladder. Data from case-control studies show higher blood BA in patients with various liver diseases, but from these designs it is unclear if the differences in BA levels are etiologic or consequential. To date no prospective studies have investigated the role of circulating BA levels in the development of HCC/GBTC, nor any potential interactions with diet, obesity and MetS. Interestingly, Vertical Sleeve Gastrectomy (VSG), an anti-obesity intervention, may alter BA profiles in some patients towards a potentially detrimental composition, but this is largely unexplored.

Project description: This project is composed of two complementary studies designed to explore the role of BA in obesity, liver function and tumourigenesis. The 1st study is a case-control study of hepatobiliary cancers (191 HCC; 266 GBTC; 457 matched controls) nested within a large prospective cohort of Franco-European populations (EPIC, >520,000 subjects) with extensive and detailed dietary/lifestyle data, body size measures and biological samples taken at baseline prior to disease development. The aim of this study is to explore associations between pre-diagnostic MetS markers and BA levels and the risk of HCC and GBTC, and to establish whether the observed associations are modulated, in part, by dietary/lifestyle factors or metabolic dysfunction.

The 2nd study is based on a clinical setting and aims to recruit 100 morbidly obese subjects undergoing VSG to compare their BA and metabolic profiles pre- to 1 year post-surgery. This study is based on observations that post-VSG BA synthesis is increased, but changes in BA composition towards possibly harmful profiles have not previously been studied. It is also hypothesized that the degree of weight loss and metabolic improvement in VSG patients may be related to pre-surgical BA profiles.

In both studies, comprehensive panel of 17 serum BA (primary, secondary, (un)-conjugated, sulphated) and metabolic biomarkers (inflammation, liver function, dyslipidemia, HbA1c, MetS indicators, hepatitis status) will be assessed using validated methods. Study 2 will also assess expression of liver FXR, a BA receptor gene. Statistical Methods: Study 1 will calculate odds ratios and 95% confidence intervals for circulating BA levels/MetS markers in relation to HCC and GBTC risk by multivariable conditional logistic regression, controlling for potential confounding variables and effect modifiers. Receiver operating characteristics (ROC) analyses will be performed to assess a combination of BA and metabolic markers with best performance to prospectively distinguish between cancer cases and controls. In study 2, GLM (repeated measures) ANOVA will be used to compare pre-/post-surgery changes in biomarkers. BA profiles from both studies, will be compared and correlations between BA and other biomarkers, lifestyle and body size measures will be assessed.

Expected results: This project is based on two related concepts. First, that lifestyle behaviours and obesity may alter gut microflora leading to changes in BA metabolism, enhancing production of specific BA known to be cancer promoting. Second, observations of increased BA levels post-VSG surgery, which may improve metabolic function, but some BA may be pro-carcinogenic over the longer term. The project will provide improved understanding of the inter-relations between BA, lifestyle behaviours and metabolic factors and the development of hepatobiliary cancers. It will also identify specific BA most strongly associated with these highly malignant cancers. The findings will contribute to the evidence base for advice on lifestyle and metabolic modifications for cancer prevention. The clinical implications are two-fold. First, the findings will provide insight as to whether BA profiles are predictive of the efficacy of VSG with potential implications in personalized medicine, and second, identified biomarker profiles may be used for more refined risk stratification for development of these cancers and subsequent closer patients' surveillance for early detection "

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo vertical sleeve gastrectomy

Exclusion Criteria:

* No liver histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo vertical sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Blood bile acids (micromols per liter) | at one year after surgery

SECONDARY OUTCOMES:
Hepatic FXR expression | At baseline
  Gene of Biliary acids Receptor

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel PERLEMUTER, MD, PhDi, Principal Investigator — Assistance Publique - Hôpitaux de Paris, Antoine Béclère Hospital
Locations (1):
- AP-HP, Antoine Béclère Hospital, Clamart, France

IPD SHARING:
Plan to Share IPD: No